CLINICAL TRIAL: NCT04491890
Title: Cross-cultural Adaptation, Evaluation and Validation of Wang Qi's Constitution of TCM Questionnaire (For Old Person)
Status: Completed | Type: Observational
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Chair Professor, Hong Kong Baptist University
Other Study IDs: HKBU JC 001
Record Dates: First submitted 2020-07-26; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Cross-cultural Adaptation, Evaluation and Validation Study of Wang Qi's Constitution in TCM Questionnaire (For Old Person)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

SUMMARY:
This is a cross-cultural adaptation, evaluation and validation study of Wang Qi's Constitution in TCM questionnaire (For Old Person) in Hong Kong to investigate the content validity, construct validity and reliability of the CTCMQ-C in Cantonese speaking Hong Kong Chinese elderly population.

DETAILED DESCRIPTION:
The study includes two steps. Firstly, translation of the questionnaire into Cantonese, followed by cross-cultural adaptation. Ten Chinese Medicine Practitioners (CMPs) and 30 patients will be recruited from the community and the outpatient clinics of Hong Kong Baptist University (HKBU) to evaluate the Constitution in TCM Questionnaire (For Old Person) (Cantonese version) (CTCMQ-C) for content validity by the cognitive debriefing interviews. The content validity indices (CVI) of clarity, relevance and appropriateness of each item of the questionnaire rated by CMPs and patients will be quantified. The interpretations of items and suggestions of rewording by the patients and CMPs will be analyzed qualitatively to identify any item of the questionnaire that is not valid for the Chinese population in Hong Kong. Secondly following the validation study, 264 patients will be recruited. A validated CTCMQ-C will then be generated and will be endorsed by expert panel to use in the subsequent cross-sectional and cohort studies to evaluate the preventive effect with Chinese Medicine approaches. The psychometric properties including construct validity by scaling assumptions, confirmatory factor analysis (CFA) and reliability of the CTMCQ-C will also be tested.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 and above;
* Hong Kong residents;
* capable of consenting and have agreed to participate.

Exclusion Criteria:

* not fulfill the above inclusion criteria;
* having serious diseases with undesirable conditions that unable to complete the survey;
* having serious mental and behavioral disorders.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: For the evaluation study of the Constitution in TCM Questionnaire (For Old Person) (Cantonese version) (CTCMQ-C), 10 Chinese Medicine Practitioners (CMPs) will be recruited from the outpatient clinics of Hong Kong Baptist University (HKBU) and 30 participants will be recruited from the community and the outpatient clinics of Hong Kong Baptist University (HKBU).
  For the validation study of the Constitution in TCM Questionnaire (For Old Person) (Cantonese version) (CTCMQ-C) (final version), 264 participants will be recruited from the community and the outpatient clinics of Hong Kong Baptist University (HKBU).
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-02-08 (Actual)

PRIMARY OUTCOMES:
To test the psychometric properties including construct validity by scaling assumptions, confirmatory factor analysis (CFA) and reliability of the Constitution in TCM Questionnaire (For Old Person) (Cantonese version) (CTCMQ-C) (final version). | 30 minutes

OTHER OUTCOMES:
To evaluate the content validity of the Constitution in TCM Questionnaire (For Old Person) (Cantonese version) (CTCMQ-C) in a Cantonese speaking Chinese elderly population in Hong Kong. | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-xiang Bian, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China